CLINICAL TRIAL: NCT03686384
Title: A Phase III, Multicenter, Randomized, Double-Blind Clinical Trial to Assess the Efficacy and Safety of SVT-15652 Otic Solution Compared to Placebo for the Treatment of Fungal Otitis Externa (Otomycosis)
Brief Title: SVT-15652 Otic Solution for the Treatment of Otomycosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Salvat (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLEAR-1
Record Dates: First submitted 2018-09-20; First posted 2018-09-26 (Actual); Results first posted 2023-01-18 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Otomycosis
MeSH Terms: conditions — Otomycosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SVT-15652 (Experimental): 1 vial twice daily
  Interventions: Drug: SVT-15652
- Placebo (Placebo Comparator): 1 vial twice daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SVT-15652 — 1 vial twice daily
  Arms: SVT-15652
Drug: Placebo — 1 vial twice daily
  Arms: Placebo

SUMMARY:
Multicenter, randomized, 2-arm parallel-group, double blind, placebo-controlled study in patients suffering from Otomycosis. This study will compare the efficacy and safety of SVT-15652 otic solution to that of Placebo, when administering one vial twice daily during 14 days.

ELIGIBILITY:
Main Inclusion Criteria:

* At least 18 years of age
* Clinical diagnosis of otomycosis in one or both ears, where topical treatment is indicated.
* Signs/symptoms of pruritus, otalgia and ear fullness.
* Debris or drainage clinically consistent with fungal infection.

Main Exclusion Criteria:

* Known bacterial otitis externa or malignant otitis externa.
* Tympanic perforation, tympanostomy tubes inserted and post mastoid surgery.
* Structural ear anomalies which may difficult the evaluation of the therapeutic response.
* Uncontrolled diabetes mellitus.
* Any infection requiring systemic antimicrobial or systemic antifungal therapy.
* Concomitant medicines that may interfere with the study evaluations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2020-02-27 (Actual); Primary Completion 2021-10-25 (Actual); Study Completion 2021-10-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Carolina Ear,Nose and Throat Clinic, Orangeburg, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The principal investigator was an otolaryngologist
Pre-assignment Details: A fungal culture was performed at baseline to know if the subject has an ear infection due to Aspergillus and/or Candida spp.
  The main efficacy population of the study was the MITT population (evaluable patients): randomized subjects who have positive baseline culture for Aspergillus and/or Candida spp.
  From the 217 subjects enrolled, 202 were treated and included in the safety population. Only 118 patients showed positive fungal culture for Aspergillus and/or Candida spp (MITT population).
Groups:
- SVT-15652: Investigational treatment
  1 vial twice daily
- Placebo: Comparator
  1 vial twice daily
Period: Overall Study
Arm/Group | SVT-15652 | Placebo
Started | 82 | 36
Completed | 75 | 21
Not Completed | 7 | 15
Not completed — Lack of Efficacy | 4 | 13
Not completed — Lost to Follow-up | 3 | 0
Not completed — Physician Decision | 0 | 1
Not completed — Took prohibited medication | 0 | 1

BASELINE CHARACTERISTICS:
Population: MITT Population: Randomized patients who had posititve baseline fungal culture for Aspergillus spp and/or Candida spp
Groups:
- Total: Total of all reporting groups
Arm/Group | SVT-15652 | Placebo | Total
Number analyzed (Participants) | 82 | 36 | 118
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.0 (17.53) | 53.4 (19.91) | 53.1 (18.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 15 | 55
  Male | 42 | 21 | 63
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 4 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 4 | 13
  White | 63 | 26 | 89
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 4 | 3 | 7
Region of Enrollment [Number; unit: participants]
  United States | 76 | 32 | 108
  Mexico | 6 | 4 | 10

OUTCOME MEASURES:

1. Primary Outcome: Therapeutical Cure (Clinical and Mycological Cure)
Description: Number and percentage of subjects with therapeutic cure
Time Frame: Test of cure on day 24
Population: MITT Population: Randomized patients who had positive baseline fungal culture for Aspergillus spp and/or Candida spp
Measure: Count of Participants; unit: Participants
Arm/Group | SVT-15652 | Placebo
Number analyzed (Participants) | 82 | 36
Participants | 48 | 10

ADVERSE EVENTS:
Time Frame: Overall study (about 4 weeks)
Description: If pre-existing signs and symptoms of otomycosis worsen during the study, this was considered a treatment failure instead of an adverse event.
  The adverse events were reviewed in the safety population which included subjects who received at least 1 dose of study medication (subjects could have positive or negative fungal culture at baseline because the results of baseline culture were not available until a few days after starting the study treatment).
Arm/Group | SVT-15652 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/134 | 0/68
Serious Adverse Events (participants affected / at risk) | 0/134 | 0/68
Other Adverse Events (participants affected / at risk) | 5/134 | 4/68
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SVT-15652 (N=134) | Placebo (N=68)
Ear pain (Ear and labyrinth disorders) | 2 (2) | 2 (2)
Headache (Nervous system disorders) | 3 (3) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication shall be expressly authorized in written by the Sponsor

DOCUMENTS (2):
  • Study Protocol (2019-10-31): https://cdn.clinicaltrials.gov/large-docs/84/NCT03686384/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-15): https://cdn.clinicaltrials.gov/large-docs/84/NCT03686384/SAP_001.pdf